CLINICAL TRIAL: NCT00085839
Title: A Randomized Phase II Study of Single Agent Erlotinib [Tarceva (TM), OSI-774] Versus Standard Chemotherapy in Patients With Previously Untreated Advanced NSCLC and a Poor Performance Status
Brief Title: Erlotinib vs. Standard Chemotherapy in Patients With Advanced Non-small Cell Lung Cancer (NSCLC) and Eastern Cooperative Oncology Group (ECOG)Performance Status (PS) 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSI-774-201
Record Dates: First submitted 2004-06-15; First posted 2004-06-17 (Estimated); Results first posted 2011-04-22 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Tarceva; NSCLC; EGFR; ECOG Performance Status 2; erlotinib; Non-Small Cell Lung Cancer; OSI-774
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Patents as Topic; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erlotinib (Experimental): Erlotinib tablets administered orally, 150 mg/day (starting dose) or 100 mg/day (reduced dose), continuous therapy
  Interventions: Drug: Tarceva (Trademark) (erlotinib HCl, OSI-774)
- Standard Chemotherapy (Active Comparator): Paclitaxel 200 mg/m^2 IV infusion over 3 hours and carboplatin AUC 6 mg/mL x min IV over 15 - 30 minutes, both given on Day 1 every 21 days for 4 cycles
  Interventions: Drug: Combination carboplatin and paclitaxel

INTERVENTIONS:
Drug: Tarceva (Trademark) (erlotinib HCl, OSI-774) — Erlotinib tablets administered orally, 150 mg/day (starting dose) or 100 mg/day (reduced dose), continuous therapy
  Arms: Erlotinib
Drug: Combination carboplatin and paclitaxel — Paclitaxel 200 mg/m^2 IV infusion over 3 hours and carboplatin AUC 6 mg/mL x min IV over 15 - 30 minutes, both given on Day 1 every 21 days for 4 cycles
  Arms: Standard Chemotherapy

SUMMARY:
The purpose of this noncomparative study is to obtain preliminary estimates of the efficacy of erlotinib and standard chemotherapy in patients with advanced, previously untreated nonsmall cell lung cancer (NSCLC) and an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 2. The study will also evaluate the safety of single-agent erlotinib in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIB or IV Nonsmall cell lung cancer (NSCLC)
* No prior chemotherapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status 2
* Clinically or radiologically measurable disease per RECIST criteria

Exclusion Criteria:

* Gastro-intestinal abnormalities
* Any concurrent anticancer therapy
* Prior treatment with epidermal growth factor receptor (EGFR) inhibitors of any kind
* Other active malignancies
* Uncontrolled brain metastases
* Severe abnormalities of the cornea
* Significant cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2004-02; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - California Cancer Care, Inc., Greenbrae, California
  - Sharp Clinical Oncology Research, San Diego, California
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Miami, Miami, Florida
  - Mount Sinai Cancer Center, Miami Beach, Florida
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - Oncology/Hematology Associates of Central Illinois, Peoria, Illinois
  - Norton Healthcare, Inc., Louisville, Kentucky
  - Maryland Hematology/Oncology Associates, Baltimore, Maryland
  - VA Sierra Nevada Health Care System, Reno, Nevada
  - Weill Medical College of Cornell University, New York, New York
  - FEK Addo, PC, Bismarck, North Dakota
  - Gabrail Cancer Center, Canton, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Charleston Hematology Oncology, Charleston, South Carolina
  - East Tennessee Oncology/Hematology, PC, Knoxville, Tennessee
  - Sarah Cannon Cancer Center, Nashville, Tennessee

REFERENCES:
- [Result] Lilenbaum R, Axelrod R, Thomas S, Dowlati A, Seigel L, Albert D, Witt K, Botkin D. Randomized phase II trial of erlotinib or standard chemotherapy in patients with advanced non-small-cell lung cancer and a performance status of 2. J Clin Oncol. 2008 Feb 20;26(6):863-9. doi: 10.1200/JCO.2007.13.2720. PMID 18281658
- See also: OSI Pharmaceuticals website — http://www.osip.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was treated 17 March 2004 and the last patient completed 19 March 2007.
Groups:
- Erlotinib: Erlotinib 150 mg/day continuous therapy
Period: Overall Study
Arm/Group | Erlotinib | Standard Chemotherapy
Started | 52 | 51
Completed | 52 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erlotinib | Standard Chemotherapy | Total
Number analyzed (Participants) | 52 | 51 | 103
Age Continuous [Median (Full Range); unit: years] | 69 [47 to 82] | 67 [47 to 84] | 68 [47 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 23 | 52
  Male | 23 | 28 | 51
Race/Ethnicity, Customized [Number; unit: participants]
  White | 35 | 33 | 68
  Black | 12 | 10 | 22
  Hispanic | 4 | 7 | 11
  Asian | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Median time until disease progression. Disease progression defined as radiological and/or symptomatic disease progression or death in absence of progression.
Time Frame: Until time of disease progression (maximum 5 months)
Population: All patients who received at least 1 dose of study drug and who had both a baseline and at least one on-treatment tumor assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib | Standard Chemotherapy
Number analyzed (Participants) | 52 | 51
months | 1.91 [1.28 to 2.69] | 3.52 [1.48 to 4.73]

2. Secondary Outcome: Overall Survival
Description: Median number of months from first study treatment until time of death
Time Frame: From first study treatment until time of death (maximum 26.8 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib | Standard Chemotherapy
Number analyzed (Participants) | 52 | 51
months | 6.57 [3.78 to 8.25] | 9.53 [7.46 to 15.54]

3. Secondary Outcome: Best Tumor Response
Description: Change in size of tumor: Complete Response (CR) = no measurable tumor; Partial Response (PR) = 30% decrease in size of measurable tumor; Stable Disease (SD) = measurable tumor size has not changed; Progressive Disease (PD) = measurable tumor 20% larger than at baseline.
Time Frame: While receiving study treatment (maximum 60 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Erlotinib | Standard Chemotherapy
Number analyzed (Participants) | 52 | 51
participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 2 | 6
  Stable Disease (SD) | 19 | 23
  Progressive Disease (PD) | 23 | 10
  Unable to Determine/Not Evaluable | 8 | 12

ADVERSE EVENTS:
Time Frame: While on study drug and 30 days after last dose
Description: Adverse events are provided regardless of causality; safety population includes patients who received at least one dose of study drug.
Arm/Group | Erlotinib | Standard Chemotherapy
Serious Adverse Events (participants affected / at risk) | 24/52 | 13/51
Other Adverse Events (participants affected / at risk) | 51/52 | 50/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=52) | Standard Chemotherapy (N=51)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Endocarditis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Pneumonia haemophilus (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Viral diarrhoea (Infections and infestations) | 1 | 0
Streptococcal infection (Infections and infestations) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiac fibrillation (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 3
Ischaemic limb pain (Vascular disorders) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0
Hypotention (Vascular disorders) | 0 | 1
Optic neuritis (Eye disorders) | 1 | 0
Death (General disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 2
Convulsion (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=52) | Standard Chemotherapy (N=51)
Nausea (Gastrointestinal disorders) | 18 | 27
Diarrhoea (Gastrointestinal disorders) | 24 | 15
Vomiting (Gastrointestinal disorders) | 12 | 15
Constipation (Gastrointestinal disorders) | 11 | 14
Dyspepsia (Gastrointestinal disorders) | 6 | 3
Stomatitis (Gastrointestinal disorders) | 6 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 5
Dysphagia (Gastrointestinal disorders) | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Dysgeusia (Gastrointestinal disorders) | 4 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 26
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 13 | 1
Rash (Skin and subcutaneous tissue disorders) | 12 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 4
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 8 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 0
Fatigue (General disorders) | 19 | 23
Oedema peripheral (General disorders) | 4 | 8
Asthenia (General disorders) | 2 | 4
Dizziness (Nervous system disorders) | 9 | 2
Headache (Nervous system disorders) | 5 | 5
Paraesthesia (Nervous system disorders) | 2 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 8
Neuropathy peripheral (Nervous system disorders) | 0 | 7
Hypoaesthesia (Nervous system disorders) | 1 | 3
Tremor (Nervous system disorders) | 3 | 1
Anorexia (Metabolism and nutrition disorders) | 18 | 16
Dehydration (Metabolism and nutrition disorders) | 4 | 4
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Weight decreased (Investigations) | 12 | 6
Insomnia (Psychiatric disorders) | 1 | 7
Anxiety (Psychiatric disorders) | 2 | 4
Confusional state (Psychiatric disorders) | 2 | 2
Depression (Psychiatric disorders) | 3 | 1
Anaemia (Blood and lymphatic system disorders) | 5 | 10
Neutropenia (Blood and lymphatic system disorders) | 0 | 4
Vision blurred (Eye disorders) | 2 | 3
Keratoconjunctivitis sicca (Eye disorders) | 2 | 2
Lacrimation increased (Eye disorders) | 3 | 1
Contusion (Injury, poisoning and procedural complications) | 4 | 1
Tachycardia (Cardiac disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less